CLINICAL TRIAL: NCT03167112
Title: A Study of Preoperative FOLFIRINOX For Potentially Curable Pancreatic Cancer
Brief Title: A Study of Administering FOLFIRINOX Before Surgery For Potentially Curable Pancreatic Cancer
Acronym: Folfirinox
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Petr Kavan (Other)
Responsible Party: Sponsor-Investigator, Petr Kavan, Dr. Petr Kavan,Director,AYA Oncology,Associate Professor,Dept. of Oncology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CODIM-MBM-17-040
Record Dates: First submitted 2017-05-14; First posted 2017-05-25 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer
Keywords: Potentially Curable; Preoperative; FOLFIRINOX
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOLFIRINOX (Experimental): Oxaliplatin, Irinotecan, Leucovorin, Fluorouracil
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin — Patients receive Oxaliplatin 85 mg/m2 over 2 hours.
  Other Names: Study regimen
Drug: Irinotecan — Oxaliplatin is followed by Irinotecan (CPT-11) 180 mg/m2 over 90 min.
  Other Names: Study regimen
Drug: Leucovorin — Oxaliplatin and Irinotecan is followed by Leucovorin (LV) 400 mg/m2 over 2 hours day1
  Other Names: Study regimen
Drug: Fluorouracil — Oxaliplatin and Irinotecan and Leucovorin is followed by Fluorouracil (5-FU) 400 mg/m2 bolus day1 and 2,400 mg/m2 46h continuous infusion.
  Other Names: Study regimen

SUMMARY:
Pancreatic cancer is a serious condition and is one of the leading cause of cancer related health problem. It is estimated that in 2016, 5,200 Canadians will be diagnosed with pancreatic cancer, and approximately 20% (1 in 5) of patients will have localized cancer (cancer that is limited to pancreas and there is no evidence of cancer in other parts of the body). Localized cancer is earlier stage of disease and surgery to remove the cancer is standard of care in this condition. However, recent scientific and clinical studies show that using the chemotherapy medication before surgery can improve the overall survival in patents with localized pancreatic cancer. One of these chemotherapy regimen is combination of fluorouracil, oxaliplatin, irinotecan, leucovorin (FOLFIRINOX) that we are going to evaluate its effect in this study.

Because of promising result of this combination in more advanced stage of pancreatic cancer, this study is going to examine its efficiency in earlier stage of pancreatic cancer (localized form). Total number of participant in this study will be 20 patients with localized form of pancreatic cancer without any evidence of cancer in other parts of the body.

Laboratory tests show that it works by slowing down the growth of cancer or may cause cancer cells to die. It is hoped that by shrinking the tumor size, the surgeon will be able to remove the cancer and improve the overall survival.

Procedures start with 2 weeks of comprehensive evaluation. Approximately 20 eligible subjects, based on this study criteria, will receive 6 treatment of this regimen every 2 weeks. Once 6 treatments have been completed, comprehensive re-evaluation procedures will be repeated, and subjects without disease progression or unacceptable toxicity will continue on their treatment based on treating team decision (surgical intervention, radiation therapy or continue FOLFIRINOX or different regimen). Patients then will follow with CT scan, blood test and physical examination every 3 months.

DETAILED DESCRIPTION:
Approximately 20% of patients present with potentially curable pancreatic cancers-resectable or borderline resectable tumors- for which surgical resection is an appropriate consideration. However, even after multimodality therapy that includes surgical resection, 5-year OS rates only reach 25% to 30% at best.

Surgical resection represents the standard of care for patients with early-stage pancreatic cancer. However, while surgical morbidity and mortality have improved over the past few decades, overall survival for pancreatic cancer has remained low. Given the increasing survival rates associated with modern chemotherapy regimens, the risks of surgery, the likelihood of R0 resection, the likelihood of subclinical metastatic disease, and the likelihood of receiving postoperative therapy (50% of patients receive post-operative chemotherapy) are our logic to evaluate preoperative chemotherapy as an alternative treatment strategy for these patients.

The main advantage of neoadjuvant chemotherapy in treating pancreatic cancer is that it significantly increases the likelihood of receiving both surgery and chemotherapy. (Winner et al., Seminars in Oncology, 2015). It is well accepted that the best results are achieved when both modalities are used. Recently, the use of FOLFIRINOX has emerged as an alternative in pancreatic cancer. A randomized trial of FOLFIRINOX versus gemcitabine in metastatic pancreatic cancer showed improved median survival from 6.8 to 11.1 months.

According to ACCORD-11 trial,FOLFIRINOX in advanced metastatic disease have demonstrated improved response rates compared with gemcitabine and other historical treatments while maintaining or improving quality of life with the median overall survival was 11.1 months FOLFIRINOX group as compared with 6.8 months in the gemcitabine group. Median progression-free survival was 6.4 months in the study regimen group and 3.3 months in the gemcitabine group, and at 6 months, 31% of the patients FOLFIRINOX group had a definitive degradation of the quality of life versus 66% in the gemcitabine group.

The role of preoperative therapy for patients with potentially curable pancreatic cancer is still unclear. The ongoing study (adjuvant gemcitabine versus neoadjuvant gemcitabine/oxaliplatin plus adjuvant gemcitabine in resectable pancreatic cancer) is a prospective randomized clinical trial that is anticipated to clarify the role of preoperative chemotherapy. However, this ongoing clinical trial does not use contemporary chemotherapy regimens with proven efficacy in higher stage settings such as FOLFIRINOX. There are only few studies evaluate this regimen in this setting.The encouraging results reported from ACCORD-11 and consequent clinical investigations prompted our group to evaluate our experience with FOLFIRINOX regimen in a selected population composed of patients with potentially curable pancreatic cancer (resectable and borderline resectable).

In this clinical trial, our primary objective is to evaluate and estimate Time to Progression (TTP). However, our secondary objectives are to determine Overall Response Rate (ORR), R0 and R1 Resection Rate, assessment of safety and toxicity associated with study regimen, and finally, to investigate Overall survival (OS).

Pre-treatment procedures start with 2 weeks of comprehensive staging evaluation. Approximately 20 eligible subjects, based on inclusion/exclusion criteria will receive study regimen for 6 treatment every 2 weeks. Once 6 treatments have been completed, comprehensive re-staging procedures will be repeated, and subjects without disease progression or unacceptable toxicity will continue on their treatment contingent upon treating team decision (surgical intervention, radiation therapy or continue chemotherapy with FOLFIRINOX or different regimen). Patients then follow with CT scan, cancer antigen 19-9 and physical examination every 3 months.

Subjects will be considered active study participants from enrollment up to survival follow-up period until documented disease progression, withdrawal of consent, lost to follow-up, or death (by any cause), whichever is earliest.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

  1. ≥ 18 years of age at the time of signing the informed consent form.
  2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures conducted.
  3. Histologically or cytologically confirmed adenocarcinoma of the pancreas.
  4. Performance status or Comorbidity condition not currently appropriate (but potentially reversible) for a major abdominal operation.

     Acceptable hematology parameters:
     1. Absolute neutrophil count (ANC) ≥ 1500 cell/mm3
     2. Platelet count ≥ 100,000/mm3 without transfusion support.
     3. Hemoglobin (Hgb) ≥ 9 g/dL

     Acceptable blood chemistry levels:
     1. Hepatic transaminases (ALT and AST) less than 2.5× the upper limits of normal (ULN)
     2. Total bilirubin level less than 1.5 × the upper limits of normal (ULN) or in patient with Biliary stenting less than 2 mg/dL
     3. Serum creatinine level less than 1.5 × the upper limits of normal (ULN) or creatinine clearance (Ccr) ≥ 40 mL/min.
     4. Alkaline phosphatase ≤ 2.5 x ULN
     5. Serum albumin > 3 g/dL

     Absence of poorly controlled comorbid conditions:
     1. Congestive heart failure (CHF)
     2. Chronic obstructive pulmonary disease (COPD)
     3. Uncontrolled diabetes mellitus (DM)
     4. Neurologic disorders (not acutely related to pancreatic cancer) or limit function
  5. Radio-graphically suspicious but not diagnostic for extra-pancreatic disease,

     1. Superior mesenteric vein and portal vein confluence that can be reconstructed even if short segment venous occlusion is present (i.e. a suitable portal vein above, and a suitable Superior mesenteric vein below the area of occlusion);
     2. Tumor abutment of the Superior mesenteric artery of ≤180⁰,
     3. Short segment encasement of the hepatic artery amenable to resection and reconstruction (this is usually at the origin of the gastroduodenal artery and reconstruction may or may not require interposition grafting with a short segment of reversed saphenous vein).
  6. Cancer antigen 19-9 level (in absence of jaundice) ≥ 100u/ml suggestive of disseminated disease.
  7. Preoperative treatment is recommended as an alternative for patients with potentially curable pancreatic cancer who meet all of the following criteria:

no clinical evidence for metastatic disease, a performance status and comorbidity condition appropriate for a major abdominal operation, no radiographic interface between primary tumor and mesenteric vasculature on imaging, an acceptable Cancer antigen 19-9 level.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Pancreatic tumors of endocrine or mixed origin.
  2. Prior anticancer therapy for pancreatic carcinoma.
  3. Presence of or history of metastatic pancreatic adenocarcinoma.
  4. Any other malignancy within 5 years prior to enrollment, with the exception of adequately treated in-situ carcinoma of the prostate (Gleason score ≤ 7), cervix, uteri, or non-melanomatous skin cancer (all treatment of which should have been completed 6 months prior to enrollment).
  5. Active bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
  6. Known infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection, or subject receiving immunosuppressive or myelo-suppressive medications that would, in the opinion of the Investigator, increase the risk of serious neutropenic complications.
  7. History of allergy or hypersensitivity to study regimen or any of their excipients.
  8. Peripheral sensory neuropathy Grade > 1.
  9. Clinically significant ascites.
  10. Plastic biliary stent. (Metal biliary stent is allowed.)
  11. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the subject's safety or the integrity of the study data. These include, but are not limited to:

      1. History of connective tissue disorders (e.g., lupus, scleroderma, arteritis nodosa)
      2. History of interstitial lung disease, slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, or multiple allergies
      3. History of the following within 6 months prior to treatment 1 Day 1: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or electrocardiogram (ECG) abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder
  12. Enrollment in any other clinical protocol or investigational study with an interventional agent or assessments that may interfere with study procedures.
  13. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
  14. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
  15. Any condition that confounds the ability to interpret data from the study.
  16. Unwillingness or inability to comply with study procedures.
  17. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Time to Progression (TTP). | Through study completion, an average of 1 year.
  Time to Progression (TTP) is defined as the time from the first cycle of chemotherapy until objective tumor progression.

SECONDARY OUTCOMES:
Overall Response Rate | Through study completion, an average of 1 year
  Overall response rate will be summarized based on RECIST V1.1
Residual (R) tumor status | Through study completion, an average of 1 year.
  The R classification is based on International Union Against Cancer (UICC).
Incidence of Treatment related Adverse Events [Safety and Tolerability] | Through study completion, an average of 1 year.
  Safety and toxicity variable is the incidence of treatment related adverse effect, serious adverse effect, laboratory abnormalities and other safety parameters.
Overall survival (OS) | Through study completion, an average of 1 year
  Overall survival indicates the interval between the first cycle of chemotherapy and the occurrence of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Kavan, MD, PhD, Principal Investigator — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Result] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Result] Katz MH, Wang H, Fleming JB, Sun CC, Hwang RF, Wolff RA, Varadhachary G, Abbruzzese JL, Crane CH, Krishnan S, Vauthey JN, Abdalla EK, Lee JE, Pisters PW, Evans DB. Long-term survival after multidisciplinary management of resected pancreatic adenocarcinoma. Ann Surg Oncol. 2009 Apr;16(4):836-47. doi: 10.1245/s10434-008-0295-2. Epub 2009 Feb 5. PMID 19194760
- [Result] Winter JM, Brennan MF, Tang LH, D'Angelica MI, Dematteo RP, Fong Y, Klimstra DS, Jarnagin WR, Allen PJ. Survival after resection of pancreatic adenocarcinoma: results from a single institution over three decades. Ann Surg Oncol. 2012 Jan;19(1):169-75. doi: 10.1245/s10434-011-1900-3. Epub 2011 Jul 15. PMID 21761104
- [Result] Katz MH, Marsh R, Herman JM, Shi Q, Collison E, Venook AP, Kindler HL, Alberts SR, Philip P, Lowy AM, Pisters PW, Posner MC, Berlin JD, Ahmad SA. Borderline resectable pancreatic cancer: need for standardization and methods for optimal clinical trial design. Ann Surg Oncol. 2013 Aug;20(8):2787-95. doi: 10.1245/s10434-013-2886-9. Epub 2013 Feb 23. PMID 23435609
- [Result] Tempero MA, Arnoletti JP, Behrman SW, Ben-Josef E, Benson AB 3rd, Casper ES, Cohen SJ, Czito B, Ellenhorn JD, Hawkins WG, Herman J, Hoffman JP, Ko A, Komanduri S, Koong A, Ma WW, Malafa MP, Merchant NB, Mulvihill SJ, Muscarella P 2nd, Nakakura EK, Obando J, Pitman MB, Sasson AR, Tally A, Thayer SP, Whiting S, Wolff RA, Wolpin BM, Freedman-Cass DA, Shead DA; National Comprehensive Cancer Networks. Pancreatic Adenocarcinoma, version 2.2012: featured updates to the NCCN Guidelines. J Natl Compr Canc Netw. 2012 Jun 1;10(6):703-13. doi: 10.6004/jnccn.2012.0073. PMID 22679115
- [Result] Oettle H, Post S, Neuhaus P, Gellert K, Langrehr J, Ridwelski K, Schramm H, Fahlke J, Zuelke C, Burkart C, Gutberlet K, Kettner E, Schmalenberg H, Weigang-Koehler K, Bechstein WO, Niedergethmann M, Schmidt-Wolf I, Roll L, Doerken B, Riess H. Adjuvant chemotherapy with gemcitabine vs observation in patients undergoing curative-intent resection of pancreatic cancer: a randomized controlled trial. JAMA. 2007 Jan 17;297(3):267-77. doi: 10.1001/jama.297.3.267. PMID 17227978
- [Result] Smeenk HG, van Eijck CH, Hop WC, Erdmann J, Tran KC, Debois M, van Cutsem E, van Dekken H, Klinkenbijl JH, Jeekel J. Long-term survival and metastatic pattern of pancreatic and periampullary cancer after adjuvant chemoradiation or observation: long-term results of EORTC trial 40891. Ann Surg. 2007 Nov;246(5):734-40. doi: 10.1097/SLA.0b013e318156eef3. PMID 17968163
- [Result] Kalser MH, Ellenberg SS. Pancreatic cancer. Adjuvant combined radiation and chemotherapy following curative resection. Arch Surg. 1985 Aug;120(8):899-903. doi: 10.1001/archsurg.1985.01390320023003. PMID 4015380
- [Result] Klinkenbijl JH, Jeekel J, Sahmoud T, van Pel R, Couvreur ML, Veenhof CH, Arnaud JP, Gonzalez DG, de Wit LT, Hennipman A, Wils J. Adjuvant radiotherapy and 5-fluorouracil after curative resection of cancer of the pancreas and periampullary region: phase III trial of the EORTC gastrointestinal tract cancer cooperative group. Ann Surg. 1999 Dec;230(6):776-82; discussion 782-4. doi: 10.1097/00000658-199912000-00006. PMID 10615932
- [Result] O'Reilly EM, Perelshteyn A, Jarnagin WR, Schattner M, Gerdes H, Capanu M, Tang LH, LaValle J, Winston C, DeMatteo RP, D'Angelica M, Kurtz RC, Abou-Alfa GK, Klimstra DS, Lowery MA, Brennan MF, Coit DG, Reidy DL, Kingham TP, Allen PJ. A single-arm, nonrandomized phase II trial of neoadjuvant gemcitabine and oxaliplatin in patients with resectable pancreas adenocarcinoma. Ann Surg. 2014 Jul;260(1):142-8. doi: 10.1097/SLA.0000000000000251. PMID 24901360
- [Result] Merkow RP, Bilimoria KY, Tomlinson JS, Paruch JL, Fleming JB, Talamonti MS, Ko CY, Bentrem DJ. Postoperative complications reduce adjuvant chemotherapy use in resectable pancreatic cancer. Ann Surg. 2014 Aug;260(2):372-7. doi: 10.1097/SLA.0000000000000378. PMID 24374509
- [Result] Wu W, He J, Cameron JL, Makary M, Soares K, Ahuja N, Rezaee N, Herman J, Zheng L, Laheru D, Choti MA, Hruban RH, Pawlik TM, Wolfgang CL, Weiss MJ. The impact of postoperative complications on the administration of adjuvant therapy following pancreaticoduodenectomy for adenocarcinoma. Ann Surg Oncol. 2014 Sep;21(9):2873-81. doi: 10.1245/s10434-014-3722-6. Epub 2014 Apr 26. PMID 24770680
- [Result] Yamada S, Fujii T, Sugimoto H, Nomoto S, Takeda S, Kodera Y, Nakao A. Aggressive surgery for borderline resectable pancreatic cancer: evaluation of National Comprehensive Cancer Network guidelines. Pancreas. 2013 Aug;42(6):1004-10. doi: 10.1097/MPA.0b013e31827b2d7c. PMID 23532000
- [Result] Bao P, Potter D, Eisenberg DP, Lenzner D, Zeh HJ, Lee Iii KK, Hughes SJ, Sanders MK, Young JL, Moser AJ. Validation of a prediction rule to maximize curative (R0) resection of early-stage pancreatic adenocarcinoma. HPB (Oxford). 2009 Nov;11(7):606-11. doi: 10.1111/j.1477-2574.2009.00110.x. PMID 20495714
- [Result] Raut CP, Tseng JF, Sun CC, Wang H, Wolff RA, Crane CH, Hwang R, Vauthey JN, Abdalla EK, Lee JE, Pisters PW, Evans DB. Impact of resection status on pattern of failure and survival after pancreaticoduodenectomy for pancreatic adenocarcinoma. Ann Surg. 2007 Jul;246(1):52-60. doi: 10.1097/01.sla.0000259391.84304.2b. PMID 17592291
- [Result] Willett CG, Lewandrowski K, Warshaw AL, Efird J, Compton CC. Resection margins in carcinoma of the head of the pancreas. Implications for radiation therapy. Ann Surg. 1993 Feb;217(2):144-8. doi: 10.1097/00000658-199302000-00008. PMID 8094952
- [Result] Davila JA, Chiao EY, Hasche JC, Petersen NJ, McGlynn KA, Shaib YH. Utilization and determinants of adjuvant therapy among older patients who receive curative surgery for pancreatic cancer. Pancreas. 2009 Jan;38(1):e18-25. doi: 10.1097/MPA.0b013e318187eb3f. PMID 18797424
- [Result] Mayo SC, Gilson MM, Herman JM, Cameron JL, Nathan H, Edil BH, Choti MA, Schulick RD, Wolfgang CL, Pawlik TM. Management of patients with pancreatic adenocarcinoma: national trends in patient selection, operative management, and use of adjuvant therapy. J Am Coll Surg. 2012 Jan;214(1):33-45. doi: 10.1016/j.jamcollsurg.2011.09.022. Epub 2011 Nov 4. PMID 22055585
- [Result] Winner M, Goff SL, Chabot JA. Neoadjuvant therapy for non-metastatic pancreatic ductal adenocarcinoma. Semin Oncol. 2015 Feb;42(1):86-97. doi: 10.1053/j.seminoncol.2014.12.008. Epub 2014 Dec 9. PMID 25726054
- [Result] Varadhachary GR, Tamm EP, Abbruzzese JL, Xiong HQ, Crane CH, Wang H, Lee JE, Pisters PW, Evans DB, Wolff RA. Borderline resectable pancreatic cancer: definitions, management, and role of preoperative therapy. Ann Surg Oncol. 2006 Aug;13(8):1035-46. doi: 10.1245/ASO.2006.08.011. Epub 2006 Jul 24. PMID 16865597
- [Result] Katz MH, Shi Q, Ahmad SA, Herman JM, Marsh Rde W, Collisson E, Schwartz L, Frankel W, Martin R, Conway W, Truty M, Kindler H, Lowy AM, Bekaii-Saab T, Philip P, Talamonti M, Cardin D, LoConte N, Shen P, Hoffman JP, Venook AP. Preoperative Modified FOLFIRINOX Treatment Followed by Capecitabine-Based Chemoradiation for Borderline Resectable Pancreatic Cancer: Alliance for Clinical Trials in Oncology Trial A021101. JAMA Surg. 2016 Aug 17;151(8):e161137. doi: 10.1001/jamasurg.2016.1137. Epub 2016 Aug 17. PMID 27275632
- [Result] Louvet C, Labianca R, Hammel P, Lledo G, Zampino MG, Andre T, Zaniboni A, Ducreux M, Aitini E, Taieb J, Faroux R, Lepere C, de Gramont A; GERCOR; GISCAD. Gemcitabine in combination with oxaliplatin compared with gemcitabine alone in locally advanced or metastatic pancreatic cancer: results of a GERCOR and GISCAD phase III trial. J Clin Oncol. 2005 May 20;23(15):3509-16. doi: 10.1200/JCO.2005.06.023. PMID 15908661
- [Result] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Result] Evans DB, Varadhachary GR, Crane CH, Sun CC, Lee JE, Pisters PW, Vauthey JN, Wang H, Cleary KR, Staerkel GA, Charnsangavej C, Lano EA, Ho L, Lenzi R, Abbruzzese JL, Wolff RA. Preoperative gemcitabine-based chemoradiation for patients with resectable adenocarcinoma of the pancreatic head. J Clin Oncol. 2008 Jul 20;26(21):3496-502. doi: 10.1200/JCO.2007.15.8634. PMID 18640930
- [Result] Varadhachary GR, Wolff RA, Crane CH, Sun CC, Lee JE, Pisters PW, Vauthey JN, Abdalla E, Wang H, Staerkel GA, Lee JH, Ross WA, Tamm EP, Bhosale PR, Krishnan S, Das P, Ho L, Xiong H, Abbruzzese JL, Evans DB. Preoperative gemcitabine and cisplatin followed by gemcitabine-based chemoradiation for resectable adenocarcinoma of the pancreatic head. J Clin Oncol. 2008 Jul 20;26(21):3487-95. doi: 10.1200/JCO.2007.15.8642. PMID 18640929
- [Result] Heinrich S, Pestalozzi B, Lesurtel M, Berrevoet F, Laurent S, Delpero JR, Raoul JL, Bachellier P, Dufour P, Moehler M, Weber A, Lang H, Rogiers X, Clavien PA. Adjuvant gemcitabine versus NEOadjuvant gemcitabine/oxaliplatin plus adjuvant gemcitabine in resectable pancreatic cancer: a randomized multicenter phase III study (NEOPAC study). BMC Cancer. 2011 Aug 10;11:346. doi: 10.1186/1471-2407-11-346. PMID 21831266
- [Result] Paniccia A, Edil BH, Schulick RD, Byers JT, Meguid C, Gajdos C, McCarter MD. Neoadjuvant FOLFIRINOX application in borderline resectable pancreatic adenocarcinoma: a retrospective cohort study. Medicine (Baltimore). 2014 Dec;93(27):e198. doi: 10.1097/MD.0000000000000198. PMID 25501072